CLINICAL TRIAL: NCT04941586
Title: Effectiveness of Pain Education in the Treatment of the Elderly With Subacromial Pain: Randomized Controlled Trial
Brief Title: Effectiveness of Pain Education Elderly Subacromial Pain
Acronym: Subacromial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rodrigo Gustavo da Silva Carvalho (Other)
Collaborators: University of Pernambuco (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Gustavo da Silva Carvalho, Clinical Professor, Universidade Federal do vale do São Francisco
Organization: Universidade Federal do vale do São Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-Subacromial
Record Dates: First submitted 2021-05-29; First posted 2021-06-28 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Shoulder Pain
Keywords: Shoulder Pain; Psychological Changes; Education in pain
MeSH Terms: conditions — Shoulder Pain | interventions — Educational Status; Musculoskeletal Manipulations; Exercise; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Experimental group: Education in Pain plus Manual Therapy plus Exercises Control group: Manual Therapy plus Exercises
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education in pain, Manual Therapy and Exercises (Experimental): The therapies will be performed by one a physical therapist with experience in rehabilitation, twice a week, lasting 60 minutes, for one month. Each therapy will last 20 minutes.
  Interventions: Other: Education in pain, Manual Therapy and Exercises
- Manual Therapy and Exercises (Active Comparator): The terapies will be performed by one a physical therapist with experience in rehabilitation, twice a week, lasting 40 minutes, for one month. Each therapy will last 20 minutes.
  Interventions: Other: Manual Therapy and Exercises

INTERVENTIONS:
Other: Education in pain, Manual Therapy and Exercises — twice a week, lasting 60 minutes, for one month
  Other Names: Education Therapy
  Arms: Education in pain, Manual Therapy and Exercises
Other: Manual Therapy and Exercises — twice a week, lasting 40 minutes, for one month
  Other Names: Manipulation Therapy; Exercises Therapy
  Arms: Manual Therapy and Exercises

SUMMARY:
Objective: To verify the effectiveness of education in pain added to other treatment modalities (manual therapy and exercises) in the outcomes of pain, functionality, depression, anxiety, stress, kinesiophobia, self-efficacy and strength.

DETAILED DESCRIPTION:
Introduction: Shoulder pain is one of the most common causes of musculoskeletal complaints found in primary care, with subacromial impact syndrome being the most common. Aging is one of the risk factors for shoulder pain. While psychological factors, which include negative beliefs about pain, catastrophization, kinesiophobia and low self-efficacy, all are related to high levels of pain and disability in the shoulder, predisposing to failure in conservative treatment. Objectives: To verify the effectiveness of pain education added to other treatment modalities (manual therapy and exercises) in the outcomes of pain, functionality, depression, anxiety, stress, kinesiophobia, self-efficacy and strength. Methodology: Randomized controlled clinical trial, which will last for one month of intervention and follow-up for three months. Primary Outcomes: Shoulder Pain and Disability Index Questionnaire that evaluates (pain and disability), Pressure Algometer (pain to pressure) and Visual Analogue Scale (pain). Secondary outcomes: Questionnaire (DASS-21), which evaluates depression, anxiety and stress, Tampa Scale (kinesiophobia), Chronic Pain Self-Efficacy Scale (Self-efficacy) and manual dynamometer that evaluates strength. 74 patients with a diagnosis of subacromial pain, of both sexes, aged between 65 and 85 years will be treated, who will be allocated into two groups: (37 patients for each group). Group A: Manual Therapy + Exercises, individual assistance, twice a week lasting 40 min. (20 min. For each therapy); Group B: Manual Therapy + Exercises + Pain Education, individual care, twice a week lasting 60 min. (20 min. For each therapy. Statistical analysis: The normality distribution will be through the Shapiro-Wilk test. For comparisons of means between and within the groups of outcomes, they will be used using the Generalized Estimation Equations and when necessary , multiple comparisons will be performed using the Bonferroni test, calculated for comparisons between the final and initial moments and initial follow-up in each group: difference in means, 95% confidence interval, effect size (d Cohen). statistical significance adopted will be 5% and the analyzes will be carried out in the statistical programs SPSS 22.0 and R 3.2.4.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 85 years old;
* Singns and symptoms of subacromial pain for at least 24 weeks;
* Medical diagnosis and ultrasound examination;
* Who do not have diseases such as: cervical radiculopathies, fractures, massive tendon ruptures, glenohumeral instabilities, dislocations and descompensated diabetes, and who have undergone surgery, infiltration or physiotherapy in the last 3 months.

Exclusion Criteria:

* Patients who do not undergo treatment in one of the groups for two consecutive sessions will be excluded from the study;
* In case the participants have any discomfort or any adverse reaction, the treatment will be suspended, after the evaluation of the evaluating researchers.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-05-29 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | change pain at four weeks and follow-up at four weeks
  Shoulder Pain and Disability Index (SPADI) (better 0- 100 worse points)
Functionality | change functionality at four weeks and follow-up at four weeks
  Shoulder Pain and Disability Index (SPADI) (better 0-100 worse points)

SECONDARY OUTCOMES:
Depression, Anxiety and Stress | change depression, anxiety and stress at four weeks and follow-up at four weeks
  Depression, Anxiety and Stress Scale (DASS-21) (better 0 - 63 worse point)
Kinesiophobia | change kinesiophobia at four weeks and follow-up at four weeks
  Tampa Scale (better 0 - 68 worse points)
Self-Efficacy | change self-efficacy at four weeks and follow-up at four weeks
  Chronic Pain Self-Efficacy Scale (worse 200 - 2.000 better points)
Muscle Strength | change muscle Strength at four weeks and follow-up at four weeks
  Hand-Held (less force worse - more strength better)
Pressure Pain | change at four weeks and follow-up at four weeks
  Pressure Algometer (an average of three applications will be the pressure-supported pain threshold)
Subjective Pain | change at four weeks and follow-up at four weeks
  Analogic Visual Scale (EVA) (better 0-10 worse points)

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Education College, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Publish Study Protocol, Randomized Controlled Trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available as of 07/18/2022.
Access Criteria: Sharing access by repository on line and journal.